CLINICAL TRIAL: NCT05081050
Title: Clinical Performance of 6-mm Short Implants Supporting Single Crowns in the Posterior Region: A 10-year Prospective Study
Brief Title: Short Implants Supporting Single Crowns in the Posterior Region
Status: Completed | Type: Observational
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CAAE 26192919.5.0000.5336
Record Dates: First submitted 2021-09-14; First posted 2021-10-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Dental Prosthesis; Dental Implants; Quality of Life
Keywords: short implants; bone loss; prosthetic complications; implant survival; bone quality; patient centred outcome measures
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 10-year Patients: Clinical and image examination to assess single crowns on short (6-mm) implants in the posterior region of the maxilla and mandible, according to functional, biological and technical variables, patient's satisfaction and quality of life.
  Interventions: Other: Only Follow-up

INTERVENTIONS:
Other: Only Follow-up — No intervention is planned.

SUMMARY:
The aim of the present project is to evaluate functional, biological and technical variables, as well as quality of life and satisfaction as indicators of long-term clinical performance of single prostheses on short implants in the posterior region with a 10-year prospective follow-up. This proposal refers to a clinical research project with a 10-year follow-up of single crowns on short implants (6 mm) in the posterior region of the maxilla and mandible. The cohort has started in 2010 through a project funded by the International Team for Implantology. The main clinical results with a 4-year follow-up showed the influence of biomechanical factors (implant/crown ratio) on short-term treatment success and increased risk over time. The sample will consist of participants from the cohort of the research project established in 2010, who received a single crown on a short implant (6-mm Standard Plus Wide Neck SLA) in the posterior region of the maxilla or mandible according to eligibility criteria and standardized clinical procedures. Data will be collected by clinical and image exams, questionnaires (for sleep bruxism, satisfaction and quality of life), recording of maximum occlusal force, measurement of perimplant bone changes, and calculation of the clinical crown-implant ratio. Data will be analyzed by descriptive and inferential statistics with survival analysis and multivariable models, if assumptions are met, at the significance level of 0.05.

DETAILED DESCRIPTION:
AIMS

General Aim:

To evaluate the clinical performance of single crowns on short (6-mm) implants in the posterior region of the maxilla and mandible, according to functional, biological and technical variables, as well as patient satisfaction and quality of life as indicators of clinical success after ten years of use.

Specific Aims: This study will

* Measure the long-term success and survival rates of short implants (6-mm) and single crowns in the posterior region, through a 10-year prospective follow-up.
* Identify risk factors for failure and complication of short implant and single crowns.
* Compare the general satisfaction and quality of life of patients with and without failures/complications.

RESEARCH DESIGN AND METHODS

Study design and sample

The study design is characterized as a cohort, prospective, observational study, as a continuation of the original clinical project established in 2010 (ITI Small Grant 688_2010: 'Risk Factors on the Prognosis of Single Short Implants in the Posterior Region - A Prospective Clinical Study'). The description and results of the 2010-cohort project have been published previously. The present protocol was approved by the University Institutional Review Board and registered in the Brazilian Ministry of Health registry 'Plataforma Brasil' (CAAE: 26192919.5.0000.5336). The study sample will consist of participants from the 2010-cohort, who were selected according to the eligibility criteria.

The 2010-cohort consisted of 20 patients who received 46 Standard Plus Wide Neck SLA (Straumann Dental Implant System, Waldenburg, Switzerland) 6-mm implants and metal-ceramic crowns cemented over SynOcta abutments (Straumann Dental Implant System, Waldenburg, Switzerland) in a private practice setting.

The patients will be recalled for a 10-year follow-up research exam and will sign a new informed consent form. Whenever possible the same instruments adopted in the first 2010-cohort study will be used for comparison purposes.

Clinical examination

Clinical data will be collected on current socio-demographic and anthropometric variables, general health, oral conditions of hard and soft tissues, occlusal status, level of oral hygiene, gingival probing, and presence of any problems with implants and prostheses.

A self-report questionnaire for diagnosis of possible bruxism will be used. The maximum occlusal force will be measured using a cross-arch compressive force transducer (Sensotec 13/2445-02, United States).

The distribution and relative force of occlusal contacts will be assessed using the T-Scan III equipment (Tekscan, United States). Patients will be asked to bite the intraoral device five times for records in centric occlusion, lateral and protrusion movements.

Patient's Perception

The patient's overall satisfaction with the treatment results will be assessed with an instrumental question: 'How satisfied are you with the results of the single crown supported by a short implant? Please rate it from zero (equal to no satisfied at all) to ten (equal to completely satisfied) on this line (10-point VAS)'.

Oral health-related quality of life will be assessed by using the OHIP-14 instrument, composed of 14 questions that cover seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, disability social, psychological disability and disability. Each question offers five alternatives: never (0), rarely (1), sometimes (2), repeatedly (3) and always (4), and the total score ranges from 0 to 56. The additive method will be used for data analysis.

Assessment of perimplant bone changes and clinical C/I ratio

Perimplant bone changes will be assessed by using periapical radiographs and cone beam computed tomography (CBCT) images for longitudinal 2-D and 3-D analyses, respectively. Periapical digital radiographs of the implants will be performed using the long cone parallelism technique. Using the computer program ImageJ version 1.3v (National Institutes of Health, Bethesda, MD, USA), the marginal bone levels in relation to the implant platform will be measured. CBCT images will be used for 3-D analysis of perimplant bone changes over time. The images will be superimposed using reference points to compute volumetric bone loss and morphological analysis of bone changes of cortical bone.

Two measurements of each outcome measure will be performed by a blind examiner with a 30-day interval for error/agreement evaluation and averaged for statistical analysis. In addition, the radiographic trabecular bone changes in density will be evaluated by means of gray levels and texture analysis variables. Longitudinal radiographic images of each implant were superimposed, and the same regions of interest were selected for measurement of gray levels statistics (mean gray levels, standard deviation and coefficient of variation) and texture parameters (correlation, contrast, entropy and angular second moment). The free software ImageJ will be used for gray levels and texture analysis by means of the GLCM Texture Tool plugin.

Clinical C/I ratio will be calculated on the periapical radiographic image: The mean bone level from the implant platform to the most coronal level of the bone-implant contact, on both mesial and distal surfaces, will be subtracted from the actual implant size to compute the clinical implant length. The clinical crown will be measured from the most coronal bone-to-implant contact point to the highest cusp point. The clinical crown value will be divided by the clinical implant value to compute the clinical C/I ratio.

Statistical analysis

Data will be analyzed by descriptive and inferential statistics at the significance level of 0.05. The success/survival estimates of implants and prostheses will be performed through survival analysis. The general satisfaction and OHIP-14 data will be analyzed to compare groups with and without complications. If preliminary assumptions are met, multiple linear regression of mixed effects models should be used. Multivariate models will be compared over time to assess possible differences in short (1 year), medium (4 years) and long (10 years) clinical follow-up periods.

Measures to Protect or Minimize Eventual Risk and Data Confidentiality

All procedures follow a protocol approved by the university IRB and biosafety standards. Data will be stored in a locked room, and access will be restricted. The PI will be legally responsible for all stages of the research development and its dissemination.

ELIGIBILITY:
The study sample will consist of participants from the 2010-cohort, who were selected according to the following eligibility criteria:

Inclusion Criteria:

* need for single implants in the posterior region of the maxilla and mandible;
* indication of 6-mm implants according to preoperative evaluation

Exclusion Criteria:

* previous problems with osseointegration failure in the region of interest;
* bone graft or use of biomaterials;
* diabetes;
* heavy tobacco use (over 10 cigarettes per day);
* immunosuppression;
* local radiation therapy;
* poor oral hygiene;
* active periodontal disease in the remaining teeth;
* cystic or neoplastic lesions;
* removable dentures in the opposing arch.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The 2010-cohort consisted of 20 patients who received 46 Standard Plus Wide Neck SLA (Straumann Dental Implant System, Waldenburg, Switzerland) 6-mm implants and metal-ceramic crowns cemented over SynOcta abutments (Straumann Dental Implant System, Waldenburg, Switzerland) in a private practice setting. The patients will be recalled for a 10-year follow-up research exam.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Ten-year Implant survival | 10-year follow-up
  Survival of short implant (6-mm) placed in the posterior region as assessed through clinical-radiographic examination at the 10-year follow-up, according to success clinical criteria, i.e., no problem that lead to implant loss or removal.
Ten-year prosthesis survival | 10-year follow-up
  Survival of single crown supported by short implant placed in the posterior region as measured through clinical-radiographic examination at the 10-year follow-up, according to success clinical criteria, i.e., no problem that lead to prosthesis loss or removal.

SECONDARY OUTCOMES:
OHIP-14 (Oral Health Impact Profile - 14) | 10-year follow-up
  Self-reported general satisfaction and oral health-related quality of life as measured by the instrument OHIP-14 (Oral Health Impact Profile - 14)
Perimplant bone change from baseline to ten years | from baseline to 10-year follow-up
  Perimplant bone change will be assessed by using radiographic images to measure the vertical bone loss from the implant platform to the most coronal level of the bone-implant contact, on both mesial and distal implant surfaces, and averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary SA Shinkai, PhD, Study Chair — Pontificia Universidade Católica do Rio Grande do Sul; Eduardo R Teixeira, PhD, Study Chair — Pontificia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD may be available to other researchers upon justified request.

REFERENCES:
- [Background] Villarinho EA, Triches DF, Alonso FR, Mezzomo LAM, Teixeira ER, Shinkai RSA. Risk factors for single crowns supported by short (6-mm) implants in the posterior region: A prospective clinical and radiographic study. Clin Implant Dent Relat Res. 2017 Aug;19(4):671-680. doi: 10.1111/cid.12494. Epub 2017 May 10. PMID 28493384
- [Background] Villarinho EA, Correia A, Vigo A, Ramos NV, Pires Vaz MA, Arai Shinkai RS. Volumetric Bone Measurement Around Dental Implants Using 3D Image Superimposition: A Methodological and Clinical Pilot Study. Int J Prosthodont. 2018 January/February;31(1):23-30. doi: 10.11607/ijp.5366. Epub 2017 Nov 16. PMID 29145529
- [Background] Triches DF, Alonso FR, Mezzomo LA, Schneider DR, Villarinho EA, Rockenbach MI, Teixeira ER, Shinkai RS. Relation between insertion torque and tactile, visual, and rescaled gray value measures of bone quality: a cross-sectional clinical study with short implants. Int J Implant Dent. 2019 Feb 11;5(1):9. doi: 10.1186/s40729-019-0158-6. PMID 30740630
- [Background] Alonso FR, Triches DF, Mezzomo LAM, Teixeira ER, Shinkai RSA. Primary and Secondary Stability of Single Short Implants. J Craniofac Surg. 2018 Sep;29(6):e548-e551. doi: 10.1097/SCS.0000000000004567. PMID 29621085
- [Background] Mezzomo LA, Miller R, Triches D, Alonso F, Shinkai RS. Meta-analysis of single crowns supported by short (<10 mm) implants in the posterior region. J Clin Periodontol. 2014 Feb;41(2):191-213. doi: 10.1111/jcpe.12180. Epub 2013 Nov 25. PMID 24266703